CLINICAL TRIAL: NCT03408288
Title: Value of an Integral Color Scale on Urine Collection Bags Versus Use of a Strip in Description of Hematuria.
Acronym: HEMAPOCHE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2017-02/AC-01
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-01

CONDITIONS: Hematuria
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses
  Interventions: Other: Hemapoche; Other: Hemastick; Other: Color description
- Urologists
  Interventions: Other: Hemapoche; Other: Hemastick; Other: Color description

INTERVENTIONS:
Other: Hemapoche — Use of Hemapoche scale to assess hematuria in reference samples
Other: Hemastick — Use of Hemastick scale to assess hematuria in reference samples
Other: Color description — Describe color of reference sample

SUMMARY:
The investigators hypothesize that incorporation of a colorimetric scale on urine collection bags to estimate degree of hematuria would allow better characterization of urine by healthcare staff thus leading to improved patient care.

ELIGIBILITY:
Inclusion Criteria:

* The participant is at least 18 year old
* Nurses recruited voluntarily in the CHU Nimes outside of the Urology department of any duration of experience
* Urologist working in the Languedoc-Roussillon region

Exclusion Criteria:

* The participant has color-blindness
* Nurse or urologist from the urology department of Nimes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses volunteering to take part in the study outside of the urology department of CHU Nimes and a panel of urologist experts
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Intra-user concordance in assessment of hematuria score measured by Hemapoche | Baseline
  Kappa coefficient
Intra-user concordance in assessment of hematuria score measured by Hemostick | Baseline
  Kappa coefficient
Intra-user concordance in assessment of hematuria described by color of urine | Baseline
  Kappa coefficient

SECONDARY OUTCOMES:
Concordance between nurses versus doctors in assessment of hematuria score measured by Hemapoche | Baseline
  Kappa coefficient
Concordance between nurses versus doctors in assessment of hematuria score measured by Hemastick | Baseline
  Kappa coefficient
Concordance between nurses versus doctors in assessment of hematuria described by color | Baseline
  Kappa coefficient
Time needed to characterize hematuria when using Hemapoche | Baseline
  Seconds (less than one minute)
Time needed to characterize hematuria when using Hemostick | Baseline
  Seconds (less than one minute)
Time needed to characterize hematuria when using color description | Baseline
  Seconds (less than one minute)
Satisfaction of medical staff in using Hemapoche medical device | Baseline
  Visual analog scale (0-10)
Usability scale of Hemapoche device according to medical staff | Baseline
  System usability scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Armand Chevrot, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France